CLINICAL TRIAL: NCT04390867
Title: A Prospective, Randomized, Cross-Over Home-Use Study of TOPS® DBS for the Treatment of Parkinson's Disease
Brief Title: Temporally Optimized Patterned Stimulation (TOPS®) Deep Brain Stimulation (DBS) for the Treatment of Parkinson's Disease
Acronym: TOPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision on June 2, 2022
Sponsor: Deep Brain Innovations LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0152
Record Dates: First submitted 2020-05-04; First posted 2020-05-18 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Random order of presentation of all three TOPS and Standard DBS in each participant
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and Outcomes Assessor blinded to DBS pattern in use
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- TOPS1 DBS (Experimental): Participants receive TOPS1 for one week if it meets screening criteria, followed by one week each of TOPS2, TOPS3, and Standard in random order.
  Interventions: Device: TOPS1 DBS; Device: TOPS2 DBS; Device: TOPS3 DBS; Device: Standard DBS
- TOPS2 DBS (Experimental): Participants receive TOPS2 for one week if it meets screening criteria, followed by one week each of TOPS1, TOPS3, and Standard in random order.
  Interventions: Device: TOPS1 DBS; Device: TOPS2 DBS; Device: TOPS3 DBS; Device: Standard DBS
- TOPS3 DBS (Experimental): Participants receive TOPS3 for one week if it meets screening criteria, followed by one week each of TOPS1, TOPS2, and Standard in random order.
  Interventions: Device: TOPS1 DBS; Device: TOPS2 DBS; Device: TOPS3 DBS; Device: Standard DBS
- Standard DBS (Active Comparator): Participants receive Standard for one week, followed by one week each of TOPS1, TOPS2, and TOPS3 in random order.
  Interventions: Device: TOPS1 DBS; Device: TOPS2 DBS; Device: TOPS3 DBS; Device: Standard DBS

INTERVENTIONS:
Device: TOPS1 DBS — TOPS1 is an investigational novel pattern of stimulation that is programmed non-invasively into an already implanted DBS system
Device: TOPS2 DBS — TOPS2 is an investigational novel pattern of stimulation that is programmed non-invasively into an already implanted DBS system
Device: TOPS3 DBS — TOPS3 is an investigational novel pattern of stimulation that is programmed non-invasively into an already implanted DBS system
Device: Standard DBS — Standard is the pattern of stimulation that is usually delivered clinically by a DBS system

SUMMARY:
This study will test newly developed stimulation settings called Temporally Optimized Patterned Stimulation or TOPS, which can be used with an already implanted deep brain stimulation system. The purpose of this study is to determine if TOPS DBS can improve Parkinson's symptoms compared to Standard DBS.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with Parkinson's disease
* Implanted with unilateral or bilateral subthalamic DBS System to treat Parkinson's disease at least 6 months prior to the study date
* Responds to DBS by having demonstrated a minimum improvement in motor score

Key Exclusion Criteria:

* Score of <24 on the Mini Mental Status Exam
* Abuses drugs or alcohol
* Pregnant
* History of significant cardiovascular, pulmonary, musculoskeletal, metabolic, or other neurological disorders (i.e. epilepsy, stroke)
* Prisoners, employees that report to investigators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
Movement Disorders Society-Unified Parkinson's Disease Rating Scale Part III Motor score - Off medication/On DBS | After 1 week treatment period using each pattern
  Average difference between the best TOPS and Standard. The MDS-UPDRS Part III is the sum of 33 scores evaluating a set of Parkinson's disease motor symptoms on a scale from 0 to 4 points. A score of 0 indicates no symptom is present and a maximum score of 4 indicates the most severe symptom. The total scale range is 0-132, where higher scores indicate more severe symptoms.
Study related adverse device effects | After 1 week treatment period using TOPS1
  Reported AEs
Study related adverse device effects | After 1 week treatment period using TOPS2
  Reported AEs
Study related adverse device effects | After 1 week treatment period using TOPS3
  Reported AEs
Study related adverse device effects | After 1 week treatment period using Standard
  Reported AEs

SECONDARY OUTCOMES:
Home Use "On Time" | During 1 week treatment period using each pattern
  Home use Parkinson's disease motor symptom diary recording On Time without dyskinesia, On Time with non-troublesome dyskinesia, On Time with troublesome dyskinesia, Off Time, and Asleep Time. Average "On Time" difference between the best TOPS and Standard
Patient Global Impression of Improvement Rating | After 1 week treatment period using each pattern
  Average difference in PGII between the best TOPS and Standard. Improvement is scored on a scale of 1 - 7 where 1 is Very Much Improved and 7 is Very Much Worse
Parkinson's Medication Use | During 1 week treatment period using each pattern
  Parkinson's medication usage recorded in home use medication diary. Average difference between the best TOPS and Standard
Rest Tremor - Off medication/On DBS | After 1 week treatment period using each pattern
  Measured using Kinesia One system. Average difference between the best TOPS and Standard
Postural Tremor - Off medication/On DBS | After 1 week treatment period using each pattern
  Measured using Kinesia One system. Average difference between the best TOPS and Standard.
Bradykinesia - Off medication/On DBS | After 1 week treatment period using each pattern
  Measured using Kinesia One system. Average difference between the best TOPS and Standard.
Type and severity of side effects of stimulation | During 1 week treatment period using each pattern
  Proportion of participants experiencing side effects recorded in home use motor symptom diary and clinic. Average difference between the best TOPS and Standard
Movement Disorders Society-Unified Parkinson's Disease Rating Scale Part III Motor score - On medication/On DBS | After 1 week treatment period using each pattern
  Average difference between the best TOPS and Standard. The MDS-UPDRS Part III is the sum of 33 scores evaluating a set of Parkinson's disease motor symptoms on a scale from 0 to 4 points. A score of 0 indicates no symptom is present and a maximum score of 4 indicates the most severe symptom. The total scale range is 0-132, where higher scores indicate more severe symptoms.
Clinical Global Impression of Improvement Rating | After 1 week treatment period using each pattern
  Average difference in CGII score between the best TOPS and Standard. Improvement is scored on a scale of 1 - 7 where 1 is Very Much Improved and 7 is Very Much Worse
Test Pattern Use Count | After 1 week treatment period using each pattern
  For each pattern, the number of subjects who go home with it and use it for the entire test period (~7-14 days) will be counted to evaluate if any patterns are more or less likely to be skipped

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No